CLINICAL TRIAL: NCT02454907
Title: The Use of Technology to Improve MS Clinical Trials and Patient Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NA_00083614
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): One kind of communication with the clinic will be used.
  Interventions: Other: Communication with the clinic
- Experimental (Experimental): A different kind of communication with the clinic will be used.
  Interventions: Other: Communication with the clinic

INTERVENTIONS:
Other: Communication with the clinic — Over the course of the study, subjects will receive brief periodic communications on their cellular phone from the doctor's office.

SUMMARY:
Many patients with multiple sclerosis (MS) experience "relapses" of disease activity during which they have increased numbness, weakness, visual problems, or other symptoms. If a person with MS has new symptoms that are concerning to them, their doctor may want to see them in the office in order to confirm that these symptoms are due to a true "relapse" of activity before starting relapse treatment. This requirement can be frustrating for patients, who may have to take time off from work or travel long distances for such unexpected doctors' visits. In this study, the investigators will use input from patients with MS and MS physicians to create a relapse questionnaire that can be used to confirm a relapse has occurred. The investigators will also evaluate if having a more direct line of communication with the provider's office improves overall patient care and satisfaction.

DETAILED DESCRIPTION:
This research is being done to study if a relapse questionnaire for people with multiple sclerosis (MS) may help more easily determine if a relapse has occurred.

A further goal of this study is to determine if receiving periodic messages from the doctor's office, as well as having the direct contact information of a person in the office, improves the care of the patients and their experience thereof.

ELIGIBILITY:
Inclusion Criteria:

* English speakers
* Relapsing-remitting MS (2010 criteria)
* Expanded Disability Status Scale (EDSS) ≤6.0
* Possession of a smartphone OR of a mobile telephone with text messaging AND an e-mail account AND web access OR willingness to be provided with, and utilize, a smartphone for the duration of the study
* In the two years before screening:

at least two relapses, OR one relapse and two new lesions (unrelated to relapse symptoms) on magnetic resonance imaging (MRI), OR RRMS (MAGNIMS 2010 criteria) onset within the past year with no exposure to disease modifying therapies (DMT)

* Patient is starting one of the following MS therapies: injectable (subcutaneous interferon beta or glatiramer acetate) or oral (fingolimod, teriflunomide, or dimethyl fumarate) therapies
* Relapse and MRI activity occurred while untreated or despite one single treatment, and no change in therapy since that activity
* Lives within 100 miles of Johns Hopkins Medical Center (Baltimore, MD)

Exclusion Criteria:

* History of DMT exposure if MAGNIMS 2010 criteria used to enroll patients with disease onset in the past year, or change in MS therapy since qualifying relapse/MRI criteria occurred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Blinded | 96 weeks
  The primary and secondary outcomes for this study are blinded.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mowry, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States